CLINICAL TRIAL: NCT00326131
Title: Pharmacokinetics and Metabolism of [14C] BMS-275183 in Patients With Advanced Cancer
Brief Title: A Phase I Study of a Single Dose of Radio-labeled BMS-275183 in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA165-017
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — taxane

INTERVENTIONS:
Drug: Oral Taxane

SUMMARY:
The first purpose of this study is to determine how the body absorbs, metabolizes, and eliminates a single dose of BMS-275183 (labeled with radioactive carbon). Secondly, to measure the levels of BMS-275183 in your blood, study the safety of the drug, and to see what effects it has on your cancer.

ELIGIBILITY:
Inclusion Criteria:

* Non-hematological malignancy that has progressed on standard therapy
* No more that 3 prior chemotherapies given for advanced cancer
* Adequate renal, hepatic and hematologic function

Exclusion Criteria:

* Uncontrolled or significant pulmonary or cardiovascular disease
* Active Brain metastases
* Inability to swallow capsules
* Serious uncontrolled medical disorder or active infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2006-04; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To assess the Pharmacokinetics, metabolism, and routes and extent of elimination of a single dose of [14C] BMS-275183 over a 10 day period.

SECONDARY OUTCOMES:
To assess the safety of a single dose of [14C] BMS-275183 followed by a therapeutic regimen of BMS-275183 administered twice weekly

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, San Antonio, Texas, United States